CLINICAL TRIAL: NCT05211869
Title: T1DTechCHW: Enhancing the Community Health Worker (CHW) Model to Promote Diabetes Technology Use in Young Adults From Underrepresented Minority Groups (YA-URMs) With Type 1 Diabetes (T1D)
Brief Title: T1DTechCHW: Enhancing the Community Health Worker Model to Promote Diabetes Technology Use in Young Adults From Underrepresented Minority Groups
Acronym: T1DTechCHW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2021-13714; R01DK132302 (NIH)
Record Dates: First submitted 2021-12-16; First posted 2022-01-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Type 1 Diabetes; Young Adult; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: 9-month randomized controlled trial in which YA-URMs will be randomized to T1D-CATCH or usual care
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be randomized after enrollment into the study using REDCap. Study staff will notify CHWs of participant assignment to the intervention arm based on REDCap. Investigators, except the PI, and outcome assessors will remain blinded to arm assignment. The PI will not be able to be blinded because they will be required to do supervision and close oversight of the CHWs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T1D-CATCH (Experimental): The CHW intervention will consist of both individual and optional group sessions with YA-URMs with T1D. In individual sessions, CHWs will provide T1D technology education, peer support, and social needs management. Over the 9-month study period, session frequency will involve weekly individual sessions based on participant technology milestones and an optional monthly CHW-led peer group support session. CHW individual and group sessions will be held via videoconferencing or in person, per participant preference and institutional COVID-19 rules.
  Interventions: Behavioral: T1D-CATCH
- Usual Care Control Condition (No Intervention): Control arm participants will receive usual primary or endocrine care at Montefiore. Usual care consists of a physician or nurse practitioner visit with review of blood sugars and treatment decisions based on provider experience. Physicians in endocrinology practices are nested within a diabetes center with access to diabetes nurse practitioners/educators, dieticians, a psychologist, and nurses. In all practices, patients are recommended to see their physician or nurse practitioner every 3 months and attend individual or group sessions.

INTERVENTIONS:
Behavioral: T1D-CATCH — As defined by the Centers for Disease Control and Prevention (CDC), a CHW is "a frontline public health worker who is a trusted member of a community or who has a thorough understanding of the community being served, and leverages this unique position to link health systems, social services, and communities". CHWs engender trust with patients by having direct community and lived experience, offering specific support and empathy that may be difficult for other diabetes care professionals to provide. In addition, CHWs have firsthand understanding of cultural barriers to traditional western healthcare and can promote patient-centered culturally-relevant care. They enhance team-based care by helping providers with extra outreach, social needs management, time-consuming tasks, and aligning patient-provider priorities.
  CHWs in this project will provide social needs assessment and management, introduction to diabetes technologies, and support for onboarding to technology.
  Arms: T1D-CATCH

SUMMARY:
The objective of this study is to test the early effects and implementation of an enhanced community health worker (CHW) model (T1D-CATCH) that encourages and supports diabetes technology use in young adults from underrepresented minority groups (YA-URMs) with type 1 diabetes (T1D). The investigators will conduct a 9-month randomized controlled trial in which YA-URMs will be randomized to T1D-CATCH or usual care. The investigators will recruit from adult and pediatric endocrinology and primary care practices in a large safety-net health system in the Bronx, New York. Our specific aims are to 1) evaluate T1D-CATCH effects on technology initiation and continued use over 6 months and 2) evaluate T1D-CATCH implementation using Proctor's Taxonomy of Implementation Outcomes: feasibility, adoption, fidelity, and cost.

DETAILED DESCRIPTION:
The study will involve a 9-month randomized control trial of usual care versus T1D-CATCH, an intervention that enhances core community health worker (CHW) service roles to support increased use of T1D technology in young adults (underrepresented minorities) (YA-URM's). Participants will be recruited from primary and specialty care practices at Montefiore Medical Center in the Bronx, New York, which is a large safety-net hospital system in one of the poorest counties in the U.S. Two young adult-aged CHWs from the Montefiore CHW program will be trained extensively per our Supporting Emerging Adults with Diabetes (SEAD) program manuals. For YA-URMs, CHWs will conduct hands-on diabetes technology education, goal-setting, peer support, and social service linkage. CHWs will also help shift insurance approval tasks away from busy providers and better align patient-provider priorities through close communication between the YA-URM and provider. Group sessions will be optional and will follow the YA-centric education curriculum developed in Dr. Agarwal's Supporting Emerging Adults with Diabetes (SEAD) program.

ELIGIBILITY:
Inclusion Criteria:

* T1D duration ≥6 months
* 18-35 years old
* Self-identified URM status: non-Hispanic Black or Hispanic
* English- or Spanish-speaking
* Not currently on a connected diabetes technology system (includes never offered, prescribed but not started within 3 months of receiving the device, discontinued, or previously refused technology)

Exclusion Criteria:

* Developmental or sensory disability interfering with study participation
* Current pregnancy
* Participation in another behavioral or diabetes technology intervention study in the past 6 months.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Technology Initiation | 6 months following intervention
  Technology use will be tracked using EMR prescriptions, self-reporting, CHW records, and device platforms and will be measured and reported as a binary variable (yes/no). Technology will include any combination of continuous glucose monitor (CGM), pump, or CGM and pump. Technology initiation will be defined as at least 1 week of first use in the 6-month period. Variables will be described using summary statistics with counts/percentages.

SECONDARY OUTCOMES:
Technology Initiation | 3 months following intervention
  Technology use will be tracked using EMR prescriptions, self-reporting, CHW records, and device platforms and will be measured and reported as a binary variable (yes/no). Technology will include any combination of continuous glucose monitor (CGM), pump, or CGM and pump. Technology use will be defined as at least 1 week of first use in the 3-month period. Variables will be described using summary statistics with counts/percentages.
Continued Technology Use - Percent Use | 9 months following intervention
  Continued technology use by study end will be determined from device platform metrics detailing days/percent time used, in addition to self-report. Per standard diabetes technology clinical trial guidelines, CGM use is defined as pump use >90% time. The percentage of time used (% used) will be summarized by study arm using basic descriptive statistics. A target of at least 90% CGM wear-time is associated with the best outcomes for glycemic control.
Continued Technology Use - Days of wear | 9 months following intervention
  Continued technology use by study end will be determined from device platform metrics detailing days/percent time used, in addition to self-report. Per standard diabetes technology clinical trial guidelines, CGM use is defined as ≥ 5/7 days wear over the 9 month period. Days of wear will be summarized study arm using basic descriptive statistics. A target of at least 5/7 days of CGM wear-time is associated with the best outcomes for glycemic control.

OTHER OUTCOMES:
Feasibility Check | 6 months (post-intervention)
  Post-intervention interviews examining intervention content, complexity, comfort, delivery, and credibility
Adoption | 9 months (post-intervention)
  Measured by recruitment logs
Adoption | 9 months (post-intervention)
  Measured by electronic medical records (EMR)
Adoption | 9 months (post-intervention)
  Measured by young adult participant consent rates
Adoption | 9 months (post-intervention)
  Measured by percentage of provider opt-in
Adoption | 9 months (post-intervention)
  Measured by CHW communications
Fidelity | Baseline
  Measured by the community health worker (CHW) dashboard
Fidelity | Baseline
  Measured by electronic medical records (EMR) to analyze session attendance
Fidelity | Baseline
  Measured by content delivery
Fidelity | 3 month mark
  Measured by community health workers (CHW) dashboard
Fidelity | 3 month mark
  Measured by CHW session recordings
Fidelity | 3 month mark
  Measured by EMR to analyze session attendance
Fidelity | 3 month mark
  Measured by content delivery
Fidelity | 3 month mark
  Measured by insurance tasks
Fidelity | 6 month mark
  Measured by CHW dashboard
Fidelity | 6 month mark
  Measured by CHW session recordings
Fidelity | 6 month mark
  Measured by EMR to analyze session attendance
Fidelity | 6 month mark
  Measured by content delivery
Fidelity | 6 month mark
  Measured by insurance tasks
Cost | 6 months (post-intervention)
  Measured by time sheets, receipts, and budget to analyze CHW salary/benefits
Cost | 6 months (post-intervention)
  Measured by time sheets, receipts, and budget to analyze CHW equipment
Cost | 6 months (post-intervention)
  Measured by time sheets, receipts, and budget to analyze CHW consumables
YA-URM Autonomy/ Competence, Social Support | Baseline
  Measured using the Healthcare Self-Determination survey
YA-URM Autonomy/ Competence, Social Support | 3 month mark
  Measured using the Healthcare Self-Determination survey
YA-URM Autonomy/ Competence, Social Support | 6 month mark
  Measured using the Healthcare Self-Determination survey
YA-URM Autonomy/ Competence, Social Support | 9 month mark
  Measured using the Healthcare Self-Determination survey
Hemoglobin A1c | Baseline
  Obtained by POC (in clinic) or laboratory (DCA Vantage)
Hemoglobin A1c | 3 month mark
  Obtained by POC (in clinic) or laboratory (DCA Vantage)
Hemoglobin A1c | 6 month mark
  Obtained by POC (in clinic) or laboratory (DCA Vantage)
Hemoglobin A1c | 9 month mark
  Obtained by POC (in clinic) or laboratory (DCA Vantage)
Quality of Life (Diabetes Distress) | Baseline
  Validated survey: Type 1 Diabetes and Life Scale - Young Adult (T1DAL-YA)
  Likert Scale: 1-5 (1= no, not at all true, 2=no, not very true, 3=sometimes true, sometimes not true, 4=yes, a little true, 5= yes, very true)
Quality of Life (Diabetes Distress) | Baseline
  Validated surveys: Problem Areas in Diabetes (PAID)
  The scores for each item are summed, then multiplied by 1.25 to generate a total score out of 100.
  * Total scores of 40 and above: severe diabetes distress
  * Individual items scored 3 or 4: moderate to severe distress to be discussed during the appointment following completion of the questionnaire.
Quality of Life (Diabetes Distress) | Baseline
  Validated survey: Diabetes Self-Management Questionnaire (DSMQ)
Quality of Life (Diabetes Distress) | Baseline
  Validated survey: Healthcare Climate Questionnaire (HCCQ)
  Likert Scale (1-7) 1= strongly disagree ---- 7= strongly agree
  Higher average scores represent a higher level of perceived autonomy support.
Quality of Life (Diabetes Distress) | 3 month follow-up
  Validated survey: Type 1 Diabetes and Life Scale - Young Adult (T1DAL-YA)
  Likert Scale: 1-5 (1= no, not at all true, 2=no, not very true, 3=sometimes true, sometimes not true, 4=yes, a little true, 5= yes, very true)
Quality of Life (Diabetes Distress) | 3 month follow-up
  Validated surveys: Problem Areas in Diabetes (PAID)
  The scores for each item are summed, then multiplied by 1.25 to generate a total score out of 100.
  * Total scores of 40 and above: severe diabetes distress
  * Individual items scored 3 or 4: moderate to severe distress to be discussed during the appointment following completion of the questionnaire.
Quality of Life (Diabetes Distress) | 3 month follow-up
  Validated survey: Diabetes Self-Management Questionnaire (DSMQ)
Quality of Life (Diabetes Distress) | 3 month follow-up
  Validated survey: Healthcare Climate Questionnaire (HCCQ)
  Likert Scale (1-7) 1= strongly disagree ---- 7= strongly agree
  Higher average scores represent a higher level of perceived autonomy support.
Quality of Life (Diabetes Distress | 6 month follow-up
  Validated survey: Type 1 Diabetes and Life Scale - Young Adult (T1DAL-YA)
  Likert Scale: 1-5 (1= no, not at all true, 2=no, not very true, 3=sometimes true, sometimes not true, 4=yes, a little true, 5= yes, very true)
Quality of Life (Diabetes Distress) | 6 month follow-up
  Validated surveys: Problem Areas in Diabetes (PAID)
  The scores for each item are summed, then multiplied by 1.25 to generate a total score out of 100.
  * Total scores of 40 and above: severe diabetes distress
  * Individual items scored 3 or 4: moderate to severe distress to be discussed during the appointment following completion of the questionnaire.
Quality of life (Diabetes Distress) | 6 month follow-up
  Validated survey: Diabetes Self-Management Questionnaire (DSMQ)
Quality of Life (Diabetes Distress) | 6 month follow-up
  Validated survey: Healthcare Climate Questionnaire (HCCQ)
  Likert Scale (1-7) 1= strongly disagree ---- 7= strongly agree
  Higher average scores represent a higher level of perceived autonomy support.

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Agarwal, MD, MPH, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal S, Schechter C, Gonzalez J, Long JA. Racial-Ethnic Disparities in Diabetes Technology use Among Young Adults with Type 1 Diabetes. Diabetes Technol Ther. 2021 Apr;23(4):306-313. doi: 10.1089/dia.2020.0338. Epub 2020 Dec 1. PMID 33155826
- [Background] Willi SM, Miller KM, DiMeglio LA, Klingensmith GJ, Simmons JH, Tamborlane WV, Nadeau KJ, Kittelsrud JM, Huckfeldt P, Beck RW, Lipman TH; T1D Exchange Clinic Network. Racial-ethnic disparities in management and outcomes among children with type 1 diabetes. Pediatrics. 2015 Mar;135(3):424-34. doi: 10.1542/peds.2014-1774. PMID 25687140
- [Background] Livingstone SJ, Levin D, Looker HC, Lindsay RS, Wild SH, Joss N, Leese G, Leslie P, McCrimmon RJ, Metcalfe W, McKnight JA, Morris AD, Pearson DW, Petrie JR, Philip S, Sattar NA, Traynor JP, Colhoun HM; Scottish Diabetes Research Network epidemiology group; Scottish Renal Registry. Estimated life expectancy in a Scottish cohort with type 1 diabetes, 2008-2010. JAMA. 2015 Jan 6;313(1):37-44. doi: 10.1001/jama.2014.16425. PMID 25562264
- [Background] Foster NC, Beck RW, Miller KM, Clements MA, Rickels MR, DiMeglio LA, Maahs DM, Tamborlane WV, Bergenstal R, Smith E, Olson BA, Garg SK. State of Type 1 Diabetes Management and Outcomes from the T1D Exchange in 2016-2018. Diabetes Technol Ther. 2019 Feb;21(2):66-72. doi: 10.1089/dia.2018.0384. Epub 2019 Jan 18. PMID 30657336
- [Background] McKergow E, Parkin L, Barson DJ, Sharples KJ, Wheeler BJ. Demographic and regional disparities in insulin pump utilization in a setting of universal funding: a New Zealand nationwide study. Acta Diabetol. 2017 Jan;54(1):63-71. doi: 10.1007/s00592-016-0912-7. Epub 2016 Sep 20. PMID 27650535
- [Background] Agarwal S, Crespo-Ramos G, Long JA, Miller VA. "I Didn't Really Have a Choice": Qualitative Analysis of Racial-Ethnic Disparities in Diabetes Technology Use Among Young Adults with Type 1 Diabetes. Diabetes Technol Ther. 2021 Sep;23(9):616-622. doi: 10.1089/dia.2021.0075. PMID 33761284
- [Background] Lai CW, Lipman TH, Willi SM, Hawkes CP. Racial and Ethnic Disparities in Rates of Continuous Glucose Monitor Initiation and Continued Use in Children With Type 1 Diabetes. Diabetes Care. 2021 Jan;44(1):255-257. doi: 10.2337/dc20-1663. Epub 2020 Nov 11. PMID 33177169
- [Background] Addala A, Auzanneau M, Miller K, Maier W, Foster N, Kapellen T, Walker A, Rosenbauer J, Maahs DM, Holl RW. A Decade of Disparities in Diabetes Technology Use and HbA1c in Pediatric Type 1 Diabetes: A Transatlantic Comparison. Diabetes Care. 2021 Jan;44(1):133-140. doi: 10.2337/dc20-0257. Epub 2020 Sep 16. PMID 32938745
- [Background] Addala A, Hanes S, Naranjo D, Maahs DM, Hood KK. Provider Implicit Bias Impacts Pediatric Type 1 Diabetes Technology Recommendations in the United States: Findings from The Gatekeeper Study. J Diabetes Sci Technol. 2021 Sep;15(5):1027-1033. doi: 10.1177/19322968211006476. Epub 2021 Apr 15. PMID 33858206
- [Background] Walker AF, Hood KK, Gurka MJ, Filipp SL, Anez-Zabala C, Cuttriss N, Haller MJ, Roque X, Naranjo D, Aulisio G, Addala A, Konopack J, Westen S, Yabut K, Mercado E, Look S, Fitzgerald B, Maizel J, Maahs DM. Barriers to Technology Use and Endocrinology Care for Underserved Communities With Type 1 Diabetes. Diabetes Care. 2021 Jul;44(7):1480-1490. doi: 10.2337/dc20-2753. Epub 2021 May 17. PMID 34001535
- [Background] Findley SE, Matos S, Hicks AL, Campbell A, Moore A, Diaz D. Building a consensus on community health workers' scope of practice: lessons from New York. Am J Public Health. 2012 Oct;102(10):1981-7. doi: 10.2105/AJPH.2011.300566. Epub 2012 Aug 16. PMID 22897548
- [Background] Saydah S, Imperatore G, Cheng Y, Geiss LS, Albright A. Disparities in Diabetes Deaths Among Children and Adolescents - United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2017 May 19;66(19):502-505. doi: 10.15585/mmwr.mm6619a4. PMID 28520705
- [Background] Walker RJ, Gebregziabher M, Martin-Harris B, Egede LE. Independent effects of socioeconomic and psychological social determinants of health on self-care and outcomes in Type 2 diabetes. Gen Hosp Psychiatry. 2014 Nov-Dec;36(6):662-8. doi: 10.1016/j.genhosppsych.2014.06.011. Epub 2014 Jul 9. PMID 25103544
- [Background] Walker RJ, Gebregziabher M, Martin-Harris B, Egede LE. Quantifying direct effects of social determinants of health on glycemic control in adults with type 2 diabetes. Diabetes Technol Ther. 2015 Feb;17(2):80-7. doi: 10.1089/dia.2014.0166. Epub 2014 Oct 31. PMID 25361382
- [Background] Berkowitz SA, Meigs JB, DeWalt D, Seligman HK, Barnard LS, Bright OJ, Schow M, Atlas SJ, Wexler DJ. Material need insecurities, control of diabetes mellitus, and use of health care resources: results of the Measuring Economic Insecurity in Diabetes study. JAMA Intern Med. 2015 Feb;175(2):257-65. doi: 10.1001/jamainternmed.2014.6888. PMID 25545780
- [Background] Berkowitz SA, Kalkhoran S, Edwards ST, Essien UR, Baggett TP. Unstable Housing and Diabetes-Related Emergency Department Visits and Hospitalization: A Nationally Representative Study of Safety-Net Clinic Patients. Diabetes Care. 2018 May;41(5):933-939. doi: 10.2337/dc17-1812. Epub 2018 Jan 4. PMID 29301822
- [Background] Hall WJ, Chapman MV, Lee KM, Merino YM, Thomas TW, Payne BK, Eng E, Day SH, Coyne-Beasley T. Implicit Racial/Ethnic Bias Among Health Care Professionals and Its Influence on Health Care Outcomes: A Systematic Review. Am J Public Health. 2015 Dec;105(12):e60-76. doi: 10.2105/AJPH.2015.302903. Epub 2015 Oct 15. PMID 26469668
- [Background] Hagiwara N, Elston Lafata J, Mezuk B, Vrana SR, Fetters MD. Detecting implicit racial bias in provider communication behaviors to reduce disparities in healthcare: Challenges, solutions, and future directions for provider communication training. Patient Educ Couns. 2019 Sep;102(9):1738-1743. doi: 10.1016/j.pec.2019.04.023. Epub 2019 Apr 19. PMID 31036330
- [Background] Franklin CM, Bernhardt JM, Lopez RP, Long-Middleton ER, Davis S. Interprofessional Teamwork and Collaboration Between Community Health Workers and Healthcare Teams: An Integrative Review. Health Serv Res Manag Epidemiol. 2015 Mar 16;2:2333392815573312. doi: 10.1177/2333392815573312. eCollection 2015 Jan-Dec. PMID 28462254
- [Background] Schaaf M, Warthin C, Freedman L, Topp SM. The community health worker as service extender, cultural broker and social change agent: a critical interpretive synthesis of roles, intent and accountability. BMJ Glob Health. 2020 Jun;5(6):e002296. doi: 10.1136/bmjgh-2020-002296. PMID 32546585
- [Background] C3 Project. The Community Health Worker Core Consensus Project (C3): Roles and Competencies. C3 Project Findings. Published 2018. Accessed April 29, 2021. https://www.c3project.org/roles-competencies
- [Background] Palmas W, March D, Darakjy S, Findley SE, Teresi J, Carrasquillo O, Luchsinger JA. Community Health Worker Interventions to Improve Glycemic Control in People with Diabetes: A Systematic Review and Meta-Analysis. J Gen Intern Med. 2015 Jul;30(7):1004-12. doi: 10.1007/s11606-015-3247-0. Epub 2015 Mar 4. PMID 25735938
- [Background] Ballard M, Westgate C, Alban R, Choudhury N, Adamjee R, Schwarz R, Bishop J, McLaughlin M, Flood D, Finnegan K, Rogers A, Olsen H, Johnson A, Palazuelos D, Schechter J. Compensation models for community health workers: Comparison of legal frameworks across five countries. J Glob Health. 2021 Feb 15;11:04010. doi: 10.7189/jogh.11.04010. PMID 33692894
- [Background] Spencer MS, Kieffer EC, Sinco B, Piatt G, Palmisano G, Hawkins J, Lebron A, Espitia N, Tang T, Funnell M, Heisler M. Outcomes at 18 Months From a Community Health Worker and Peer Leader Diabetes Self-Management Program for Latino Adults. Diabetes Care. 2018 Jul;41(7):1414-1422. doi: 10.2337/dc17-0978. Epub 2018 Apr 27. PMID 29703724

DOCUMENTS (1):
  • Informed Consent Form (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT05211869/ICF_002.pdf